CLINICAL TRIAL: NCT04476758
Title: Immune Profiles in CF Fungal Infection
Status: Completed | Type: Observational
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: University of Colorado, Denver (Other)
Responsible Party: Principal Investigator, Thomas Spencer Poore, Assistant Professor, University of Alabama at Birmingham
Other Study IDs: 20-0099; POORE20D0 (Other Grant/Funding Number: Cystic Fibrosis Foundation)
Record Dates: First submitted 2020-07-08; First posted 2020-07-20 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-07

CONDITIONS: Cystic Fibrosis; Fungal Infection; Allergic Bronchopulmonary Aspergillosis
Keywords: Fungal Infection; Th2 Inflammation; Cystic Fibrosis; Fungal allergy; Allergic Bronchopulmonary Aspergillosis
MeSH Terms: conditions — Cystic Fibrosis; Mycoses; Aspergillosis, Allergic Bronchopulmonary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Sputum and serum from subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Fungal Infection Group: Have had a fungal species isolated from sputum and/or BAL culture on >= 2 separate occasions in the 18 months preceding study visit and do not have a diagnosis of ABPA (N=10).
- Control Group: Have never previously isolated fungus from sputum, BAL, or OP swab (N=10).
- ABPA Group: Previous diagnosis of ABPA as defined by CFF guidelines, regardless of the amount of fungal infection or history thereof.
  • ABPA Minimum diagnostic criteria per CFF: Acute or subacute deterioration, total serum IgE > 500 IU per mL, immediate cutaneous reactivity to Aspergillus or in vitro IgE antibody to A. fumigatus, and either a new or recent chest imaging change that has not responded to antibiotics and standard physiotherapy OR precipitin to A. fumigatus or IgG antibody to A. fumigatus1 (N=5). Culture positive sputum is not required for ABPA diagnosis and is not taken into account for the diagnosis per CFF guidelines.

SUMMARY:
This study is investigating the role of allergic (Th2) inflammation in patients with Cystic Fibrosis (CF) and history of fungal infection and/or Allergic Bronchopulmonary Aspergillosis. Little is known about fungal infection in CF and conflicting results exist on whether this results in worse lung function over time. There is concern that persistent fungal infection can result in worse clinical outcome measures in patients with CF. Also, it is unclear how ABPA develops, but may be related to the amount of fungus a patient with CF is infected with. This study looks at inflammatory patterns and allergic responses to fungal elements to help identify biomarkers and signs of allergic disease in fungally infected patients with CF.

DETAILED DESCRIPTION:
While bacteria are predominant agents in CF lung disease, fungi are often isolated in both sputum and bronchoalveolar lavage fluid (BAL), yet their role in CF is not fully understood. Fungal infection in CF has a wide spectrum of presentations, varying from transient detection to persistent infection, acute fungal bronchitis with resulting pulmonary exacerbation, sensitization to fungal allergens, and allergic bronchopulmonary aspergillosis (ABPA). While there are clinical guidelines for the diagnosis and treatment of ABPA in patients with CF, there are few guidelines and recommendations regarding monitoring, clinical care, and antifungal treatment in the various presentations of CF fungal disease; further, the clinical impact of fungi without ABPA is poorly understood. While inflammation in CF is classically considered a neutrophil and macrophage driven process (Th1), eosinophils and allergic cytokines (Th2) have been shown to be elevated in the presence of fungal disease in both clinical and animal CF studies. Studies have also shown decreased lung function (e.g. percent predicted forced expiratory volume in one second, ppFEV1) in individuals with frequent fungal detection in their sputum, and associations with Pseudomonas infection and use of antimicrobials. Adults with CF are also more prone to fungal sensitization when compared to non-CF patients as well as having higher rates of allergic rhinitis and atopy. In a retrospective study performed at our center, we found that children with intermittent or chronic fungal infections experienced more rapid decline in lung function compared to those without fungal infections regardless of ABPA status (see preliminary data). Understanding whether fungal infections are driven by an allergic (Th2) inflammatory process may alter treatment approaches by utilizing steroids and antifungal therapies more readily in patients with fungal infection to combat lung function decline. Limited studies have investigated the frequency of allergic sensitization to fungal pathogens in individuals with CF, the frequency of allergic sensitization in the pediatric CF population in general, and the unique inflammatory profiles and phenotypes of CF fungal infections, both in the sputum and the serum.

Hypothesis: We hypothesize that children with CF and fungal infections without ABPA will have elevated allergic inflammatory profiles and increased sensitization to fungal elements compared to those without fungal infection.

Specific Aim 1: Compare Th2 inflammation in patients with and without fungal infections in patients with CF and to those with ABPA.

* Approach: We will obtain serum and sputum samples from 25 patients with either (1) fungal infection without ABPA, n=10 (defined as ≥ two positive fungal cultures in prior 18 months), (2) no fungal infection, n=10, and (3) ABPA, n=5, and measure specific sputum and serum cytokine measurements to evaluate Th2 and Th1 inflammatory pathways.
* Biomarkers measured: Eosinophilic cationic protein (ECP), Interleukin-4 (IL4), Interleukin-5 (IL5), Interleukin-10 (IL10), Interleukin-13 (IL13), and eosinophil count in both serum and sputum.
* Expected outcome: Individuals with fungal infection without APBA will have elevated Th2 markers of inflammation compared to those with no fungal infection. We will also compare to those with ABPA as a separate control group. We will also measure Th1 markers to be used as a reference to previously established inflammatory profiles seen in CF, seeing if those with fungal disease deviate towards a more Th2 driven process.

Specific Aim 2: Investigate allergic sensitization to fungal elements in patients with CF fungal infection without ABPA compared to those without fungal infection and to those with ABPA.

* Approach: We will measure total IgE and serum ImmunoCAP testing of specific IgE levels to fungal proteins of various species (Aspergillus, Candida, etc). to determine fungal sensitization. We will also survey patients regarding environmental exposures to explore relationships with allergic sensitization.
* Expected outcome: Individuals with fungal infection without ABPA will be more likely to show allergic sensitization to fungal elements when compared to those with no fungal infection.

The results of this study will help characterize the inflammatory profile associated with CF fungal infections contributing to the understanding of both the infectious and allergic nature of disease in the CF population. From this, the contribution to both the pathophysiology and clinical characteristics of CF fungal infections will serve as a step towards understanding management options, care guidelines, and disease progression for this unique set of hard to treat organisms.

Recruitment: We propose to recruit 25 patients with CF aged between 8 and 25 years who agree to participate in this cross-sectional study looking at the immune system characteristics of fungal infection and ABPA. We plan to screen individuals coming to their routine CF clinic and approach them regarding their interest in participating in this study. From this, we will explain the concept, hypothesis, and procedures involved with intent to schedule them for a research visit.

Patient Selection: Patients will be recruited from the CF Center at CHCO by study investigators or qualified research coordinators at the time of a routine clinic visit.

Study Visit: We plan to prospectively recruit 25 subjects with CF during a period of clinical stability. Subjects will have one research clinic visit that will coincide with their clinic visit at CHCO Pulmonary Clinic facilities. The following diagnostic information will be entered onto Case Report Forms: demographic information, diagnostic history and mutations, CF-related co-morbidities, historic microbiology results including fungal culture results, medications including modulator therapy and long-term antibiotic regimens, previous allergy testing, diagnostic criteria for ABPA (if applicable). We will also utilize historical clinical data from the medical record to establish other co-morbidities, lung function trends and baseline, history of other bacterial infections, history of allergy diagnoses, and other pertinent medical history and diagnostic testing (ie previous CT scan results, previous blood work, etc.). The following evaluations will be performed :

* Historical data in the medical record. Examples include Co-morbid diagnoses related to CF (such as but not limited to CF related diabetes, CF liver disease, asthma, etc), previous blood work (such as but not limited to serum IgE levels, previous allergy testing, bronchoscopy data and lavage studies, routine and urgent/admission CF labs, etc), previous spirometery and lung function data, previous nutritional and growth data (BMI, vitamin levels, etc), previous microbiology and culture data, etc.
* BMI measurements obtained from regular CF clinic visit
* Height and weight to be obtained and subsequently calculated.
* Pulmonary function testing obtained from regular CF clinic visit. Spirometry will be performed according to American Thoracic Society criteria, while absolute values will be converted to percent predicted using the Global Lung Function initiative reference equations34.
* Sputum collection. Spontaneously expectorated sputum will be used as possible.This will be collected at home by the patient following a routine respiratory airway clearance regimen within 12 hours of clinic visit. The sample will be placed in a mailed specimen cup and placed on ice and brought to the clinic visit. If sputum is not able to be expectorated prior to visit, we will attempt to utilize remaining sputum expectorated that is not used for clinical needs for further analysis and storage. Sputum may be collected by sputum induction according to the current CFF Therapeutics Development Network standard operating procedure if 1) unable to expectorate, (2) patient meets clinical criteria for sputum induction and (3) clinic is able to perform research induced sputum based on current COVID-19 guidelines to ensure safety of team member and adequate PPE supply.

For safety reasons, the induction procedures will only be performed for subjects who meet the following criteria on the day of the induction: FEV1 ≥ 30% predicted, No history of > 5 mL hemoptysis within 48 hours prior to the visit, Able to tolerate the sputum induction procedure. Of note, there is little significant difference in specimen quality for analysis between expectorated and induced sputum. Markers to be tested as previously described above.

* Environmental fungal exposure questionnaire. Will be performed prior to finish of clinic visit. This questionnaire in entirety is a validated questionnaire used by Dr. Andy Liu. Given time constraints for study participants, we are using a modified questionnaire focused on questions of interested to this study (e.g. pertaining to fungal exposure). This has not been validated but may provide important information in this pilot study for future research
* Serum collection. Peripheral venous blood draw will be performed by certified individual using appropriate sterile technique by the CTRC. Samples will be labeled per research protocol standards. Markers to be tested described above.

  * All sputum samples to be banked and saved for potential microbiome, mycobiome and transcriptome analysis, assessing gene expressions unique to various inflammatory pathways.

Sample Size Estimates: Power and sample size for the study proposal is fixed due to the expected number of eligible patients to be recruited into this pilot study during the study window. Based on preliminary data and the described definitions of types of infection, investigators anticipate that over a 1-year recruitment window they will be able to enroll approximately 10 individuals with no fungal infection, 10 patients with a fungal infection but not ABPA and 5 with ABPA. The primary analysis plan focuses on the description and comparison of key plasma and sputum measures described in Table 3. Power analysis provides the detectable effect sizes when comparing the control arm (no fungal infection) to either the non-ABPA group or the ABPA group. Calculations are based on a power of 80% and Type I error rate of 0.05 for two-sided two-sample equal-variance t-test conducted in PASS version 15 statistical software (2). Group sample sizes of 10 and 5 in the fungal infection groups achieve 80% power to reject the null hypothesis of zero effect size when the population effect size is 1.36 and 1.66 respectively. Thus, the study is powered at 80% to detect a difference in the mean markers to be measured greater than 1.66 and 1.32 standard deviations. Given limited data in the literature regarding Th2 markers in CF, we are basing these calculations off of deviations from a mean for the multiple Th2 markers we are testing.

Data Collection and Storage: All subjects will be de-identified upon study sample collection and stored with a master key. There will be limited access to this information with the PI and only essential research staff able to monitor and view the data. All hardcopy source documents will be kept in a locked file cabinet in the CF research team's storage facilities. Additionally, to further ensure data integrity, data for this study will be stored in Research Electronic Data Capture system (REDCap), which will allow limited access to only essential personal. REDCap enables in-line validation to minimize transcription errors and provides real-time notifications of data submission and allows immediate central monitoring and feedback. Access to data requires an encrypted secure socket layer (SSL) connection and changes are logged by user ID, time stamp and project. Databases are backed up frequently.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CF per CFF guidelines and followed at Children's Hospital Colorado (CHCO) CF Center
* Meets criteria of only one fungal group (described below)
* Clinical stability without any change acute antibiotic regimen in the past 14 days
* Clinical stability without any use for acute NSAID or oral steroids in past 14 days
* Individuals with other co-morbid conditions related to and unrelated to CF, including but not limited to CF related diabetes, CF related liver disease, asthma, etc.

Exclusion Criteria:

* History of Burkholderia sp. or Non-tuberculosis Mycobacterium
* Comorbid or health contraindication to induced sputum treatment or blood draw

Ages: 8 Years to 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: Pediatric to young adult patients with CF followed at Children's Hospital Colorado. Patients must meet inclusion/exclusion criteria and fit into one of the three groups described.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2021-02-10 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Difference in Th2 Sputum Markers | Day 1
  Difference in sputum Th2 biomarkers (ECP, IL4, IL5, IL10, IL13, and eosinophil count) in patients with CF with fungal infection with expected elevation of sputum Th2 biomarkers in patients with CF and ABPA compared to those without fungal infection and without ABPA.

SECONDARY OUTCOMES:
Other markers of fungal inflammation and allergic reaction in patients with CF | Day 1
  * Serum Th2 biomarkers in patients with fungal infection and ABPA (Table 3).
  * Serum Th1 biomarkers in patients with fungal infection and ABPA (Table 3).
  * Serum sensitization markers to fungal allergens in patients with fungal infection and ABPA (Table 4).
  * Baseline and historic lung function, historical comorbid diagnoses and BMI measurements in patients with fungal infection and ABPA.
  * Environmental factors that are possibly related to fungal infection and ABPA in patients with CF.
  * Immune profile: A profile of each group will be based upon their findings of each set of biomarkers: Th1, Th2, mold allergy panel, and systemic markers of inflammation. Based upon findings in each of these categories (elevated, depressed), we will be able to formulate a profile based upon the type of marker/inflammatory pathway.

OTHER OUTCOMES:
Biobanking of specimens | Day 1
  Banking of both sputum and serum to potentially utilize microbiome and transcriptome techniques for further immunotyping and infection characterization.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas S Poore, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Childrens Hospital Colorado, Highlands Ranch, Colorado, United States

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT04476758/Prot_SAP_000.pdf
  • Informed Consent Form (2020-06-10): https://cdn.clinicaltrials.gov/large-docs/58/NCT04476758/ICF_001.pdf